CLINICAL TRIAL: NCT03350061
Title: Restoration of Sensations From the Lost Limb to Amputees for Fall Avoidance, Regular Walking, Phantom Limb Pain Diminishment and Embodiment of Prosthesis
Brief Title: Prosthesis With Sensations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Centre of Serbia (Other)
Collaborators: Axonic (Unknown); SensArs Neuroprosthetics Sarl (Industry); Institut für Mikrosystemtechnik (IMTEK), Albert-Ludwigs-Universität Freiburg (Unknown); Ripple LLC (Unknown); Össur hf (Unknown)
Responsible Party: Principal Investigator, Francesco Petrini, President, SensArs Neuroprosthetics Sarl
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Osecaj Opet
Record Dates: First submitted 2017-11-12; First posted 2017-11-22 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Amputation; Phantom Limb Pain; Sensory Deficit
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SENSY benefit (Experimental): Sensory feedback elicited by intraneural stimulation will be provided by SENSY with and without the leg prosthesis to improve walking ability, increase embodiment, and reduce metabolic cost, cognitive load and phantom pain.
  Interventions: Device: SENSY

INTERVENTIONS:
Device: SENSY — The sensory feedback will be delivered by SENSY with or without the leg prosthesis. Benefits connected to the stimulation of sensory nerves will be assessed.

SUMMARY:
Lower limb amputees suffer complete lack of sensory feedback of current available prostheses, which excludes the central nervous system from the correct sensory-motor integration. It causes serious problems as: falls due to unexpected perturbations, asymmetric walking, low mobility, higher power consumption, feeling the prosthesis as a foreign body, high cognitive burden, and phantom limb pain occurrence.

Investigators will provide amputees with a prosthesis restoring sensory feedback and will assess its benefits on the users.

DETAILED DESCRIPTION:
The clinical investigation described here aims at evaluating the benefit of a lower limb prosthesis providing sensory feedback (bidirectional prosthesis), in selected transfemoral amputees. The device is constituted by i) Rheo Knee XC, Pro Flex foot and customized socket/liner structure from OSSUR. Rheo Knee embedded already an encoder coupled with a Bluetooth unit, which is used to make communication with devices external to the knee itself; ii) nerve stimulating system constituted by implantable intraneural electrodes from IMTEK, iii) an external neurostimulator from AXONIC, and iv) sensorized sole from SensArs Neuroprosthetics to apply under the prosthetic foot and driving the stimulating system. The readout of the sensorized insole are transmitted via Bluetooth, together with the encoder readout, to an external controller, which transduces it in parameters of stimulation. These parameters are sent to the stimulator, which injects current into the intraneural electrodes. As final result, the subject perceives sensory feedback from the prosthesis when using it.

Investigators call SENSY the sensory feedback restoration system. The subjects will use the prosthesis with and without sensory feedback to execute walking tasks. The average change of kinematics (including falls), metabolic cost, embodiment, and cognitive burden (EEG) when intraneural stimulation is provided will be compared to the case in which there is no sensory feedback. Standard clinical tests (as PEQ and CB&MS) will be executed with and without sensory feedback. Also, when the subjects will report attacks of phantom pain, they will undergo a 10-minutes-stimulation session. Only stimulation without prosthesis is used in this intervention.

Finally, imaging of the cortical activity will be executed through functional magnetic resonance imaging (fMRI). This procedure will be only observational since no prosthesis or sensory feedback will be used by the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Uni-lateral transfemoral amputation above the knee level
* Other treatments for phantom limb pain should have been tried with poor results
* The subject should experience phantom limb pain at a level of 6 or higher measured on on a visual analog scale (VAS) ranging from 0-10
* Phantom limb pain should be experienced at least once a week
* The subject should be in a chronic and stable phase, and the stump should have healed
* The subject should otherwise be healthy and able to carry out the experiment
* If pain medication is used it will be acceptable that the person continues to use the medication

Exclusion Criteria:

* Cognitive impairment
* Pregnancy
* Prior or current psychological diseases such as borderline, schizophrenia, depression or maniodepression
* Acquired brain injury with residual impairment
* Prior neurological or musculoskeletal diseases
* History of or active substance abuse disorder
* Excessive sensitivity to electrical stimulation with surface electrodes
* Persons with fear for electrical stimulation, pain cannot participate
* Persons that are hypersensitive to electrical stimulation and experience the stimulation as unpleasant cannot participate
* Since the protocol includes MRI scanning of the brain, persons that may feel claustrophobic cannot participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-11-12 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Impact of SENSY on mobility | within 3 months post implant
  Demonstration of statistically relevant increase of kinematic walking speed (distance/minute) during the execution of tests involving the use of the prosthesis with intraneural stimulation compared to without the stimulation (e.g. climbing and descending stairs, tandem walking, walking on an outdoor surface).
Impact of SENSY on falls avoidance | within 3 months post implant
  Demonstration of statistically relevant decrease of falls during the execution of tests involving the use of the prosthesis with intraneural stimulation compared to without the stimulation (e.g. walking on a surface with obstacles).
Impact of SENSY on metabolic consumption | within 3 months post implant
  Demonstration of statistically relevant decrease of metabolic cost during the execution of tests involving the use of the prosthesis with intraneural stimulation compared to without the stimulation (e.g. walking on the treadmill and walking on an outdoor surface). Metabolic cost is measured as volume of oxygen (VO2) consumption (mLO2/kg/meter).
Incidence of all serious adverse events concerning SENSY | within 3 months post implant
  Incidence of all serious adverse events, including Serious Adverse Events, Serious Adverse Device Events, and Unanticipated (Serious) Adverse Device Events from the time of consent through 3 months post implant.

SECONDARY OUTCOMES:
Impact of SENSY on phantom pain: neuropathic pain symptom inventory score | within 3 months post implant
  Demonstration of statistically relevant reduction in neuropathic pain symptom inventory (NPSI) pain score (0-100) from pre-treatment to post-treatment (10-minutes stimulation session is the treatment).
Impact of SENSY on phantom pain: visual analog scale score | within 3 months post implant
  Demonstration of statistically relevant reduction in visual analog scale (VAS) pain score (0-10) from pre-treatment to post-treatment (10-minutes stimulation session is the treatment).
Impact of SENSY on phantom pain before and after the implant of SENSY: NPSI score | until up to 3 months post explant
  Average change in NPSI pain score among 1 day pre-implant, 1 day pre-explant, 1.5 and 3 months after the explant.
Impact of SENSY on phantom pain before and after the implant of SENSY: VAS score | until up to 3 months post explant
  Average change in VAS pain score among 1 day pre-implant, 1 day pre-explant, 1.5 and 3 months after the explant.
Impact of SENSY on embodiment (perception of the prosthesis as part of the body): questionnaires | within 3 months post implant
  Average change of embodiment (measured through questionnaires) after use of the prosthesis with and without intraneural stimulation.
Impact of SENSY on embodiment (perception of the prosthesis as part of the body): proprioceptive drift | within 3 months post implant
  Average change of embodiment (measured through proprioceptive drift) after use of the prosthesis with and without intraneural stimulation.
Impact of SENSY on cognitive effort | within 3 months post implant
  Average change of cortical burden (measured as electroencephalography (EEG) activity) during use of the prosthesis with and without intraneural stimulation.
Impact of SENSY on cortical plasticity | within 3 months post explant
  Average cortical reorganization measured through functional Magnetic Resonance Imaging between after the implant and after the explant.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Lešić, Prof, Study Director — Clinical center of Serbia
Locations (1):
- Clinical center of Serbia, Belgrade, RS, Serbia

REFERENCES:
- [Derived] Valle G, Katic Secerovic N, Eggemann D, Gorskii O, Pavlova N, Petrini FM, Cvancara P, Stieglitz T, Musienko P, Bumbasirevic M, Raspopovic S. Biomimetic computer-to-brain communication enhancing naturalistic touch sensations via peripheral nerve stimulation. Nat Commun. 2024 Feb 20;15(1):1151. doi: 10.1038/s41467-024-45190-6. PMID 38378671
- [Derived] Petrusic I, Valle G, Dakovic M, Damjanovic D, Bumbasirevic M, Raspopovic S. Plastic changes in the brain after a neuro-prosthetic leg use. Clin Neurophysiol. 2022 Jun;138:186-188. doi: 10.1016/j.clinph.2022.04.001. Epub 2022 Apr 9. No abstract available. PMID 35461007
- [Derived] Preatoni G, Valle G, Petrini FM, Raspopovic S. Lightening the Perceived Prosthesis Weight with Neural Embodiment Promoted by Sensory Feedback. Curr Biol. 2021 Mar 8;31(5):1065-1071.e4. doi: 10.1016/j.cub.2020.11.069. Epub 2021 Jan 7. PMID 33417885
- [Derived] Petrini FM, Bumbasirevic M, Valle G, Ilic V, Mijovic P, Cvancara P, Barberi F, Katic N, Bortolotti D, Andreu D, Lechler K, Lesic A, Mazic S, Mijovic B, Guiraud D, Stieglitz T, Alexandersson A, Micera S, Raspopovic S. Sensory feedback restoration in leg amputees improves walking speed, metabolic cost and phantom pain. Nat Med. 2019 Sep;25(9):1356-1363. doi: 10.1038/s41591-019-0567-3. Epub 2019 Sep 9. PMID 31501600